CLINICAL TRIAL: NCT00645567
Title: Evaluation of Transfer Technologies to Preserve Shoulder Function in SCI
Brief Title: Biomechanics of Wheelchair Transfers
Status: Completed | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: B6103-R
Record Dates: First submitted 2008-03-19; First posted 2008-03-27 (Estimated); Results first posted 2017-04-07 (Actual); Last update posted 2017-04-07 (Actual); Status verified 2017-04

CONDITIONS: Spinal Cord Injury
Keywords: Biomechanics; Ergonomics; Spinal Cord Injury; Pain; Shoulder
MeSH Terms: conditions — Spinal Cord Injuries; Pain

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Unassisted manual transfer: this group will use no additional aid in transfer.
  Interventions: Device: Unassisted Manual Transfer
- Standard sliding board transfer: The standard transfer board is a flat surface board designed to bridge the gap that exists with transfers from wheelchair to vehicle and/or other horizontally displaced seating surfaces.
  Interventions: Device: Standard Transfer Board
- Glide n' Go Lift: The Glide n' Go lift is a flip down power list seat that enables the person to enter and exit the vehicle by lifting them from their wheelchair up tot eh vehicle seat that they can make an easy transfer into the vehicle. Trunk stability may be required to successfully use the device.
  Interventions: Device: Glide n' Go
- Easy Reach lift: The Easy Reach lift seat allows the vehicles original seat to swivel out of the vehicle and lower to wheelchair height. the chair extends far from the vehicle to provide access for a safe, easy transfer.
  Interventions: Device: Easy Reach lift
- Ryno lift: The Ryno lift is an under-vehicle list (UVL) system. Using this lift, the wheelchair user is raised into the vehicle cab using independent controls and can then maneuver into a convenient position in the cab. The wheelchair is locked down and the lift stored beneath the vehicle chassis. This technology eliminated the need to store and retrieve a wheelchair during transit.
  Interventions: Device: Ryno lift

INTERVENTIONS:
Device: Unassisted Manual Transfer — No device assistance
  Groups: Unassisted manual transfer
Device: Standard Transfer Board — Flat surface board
  Groups: Standard sliding board transfer
Device: Glide n' Go — Flip down power lift chair
  Groups: Glide n' Go Lift
Device: Easy Reach lift — Original chair is converted to a chair that swivels out of the vehicle and lowers to wheelchair height
  Groups: Easy Reach lift
Device: Ryno lift — Lift for the wheelchair
  Groups: Ryno lift

SUMMARY:
This is a laboratory-based study to evaluate the risk of shoulder injury associated with transfers between wheelchair and vehicle in persons with spinal cord injury. Four new devices will be compared against an unassisted transfer.

DETAILED DESCRIPTION:
Specific Aims:

The purpose of this 3 year laboratory-based randomized crossover study is to evaluate the ergonomic effectiveness of four wheelchair/vehicle transfer assistive devices, including (1) standard transfer board, (2) Glide n' Go, ( 3) Easy Reach Lift, and (4) Ryno Lift, and to compare them to an unassisted manual transfer. We have targeted persons with paraplegia (level of injury T2-L5) to standardize physical capabilities. Our research questions are:

1. Evaluate the impact of vehicle/wheelchair transfers on objective measures of shoulder kinematics, kinetics, and muscle activity, for each of the participants.
2. Evaluate the impact of vehicle/wheelchair transfers on subjective measures of shoulder pain, spasticity, perceived comfort, ease, efficiency, and safety.
3. Examine the effects of covariates (patient characteristics, SCI characteristics and pain) on both objective and subjective outcome measures.

Background:

Upper limb pain and injury are highly prevalent in persons with a spinal cord injury (SCI) who use a manual wheelchair for mobility. Historically, persons with paraplegia did not long survive the trauma of their injury, but with advances in medicine and emergency services, persons with SCI now have a life expectancy approaching that of the general population. For persons with paraplegia, paralysis of the lower limbs necessitates an over reliance on the upper limbs for performing wheelchair propulsion, transfers in/out of the wheelchair, and other mobility-related tasks. Many years of overuse of the upper extremities leads to an increased incidence of pain and cumulative trauma to the shoulders, elbows and wrists. Over 50% of persons with SCI have upper extremity pain; rotator cuff tears have been reported in 59-73%; and 40% have clinical evidence of carpal tunnel syndrome. Upper extremity deterioration following years of compensating for the lack of functional lower limbs in addition to their usual loading reduces quality of life, function, independence, and even life expectancy following SCI. The two most stressful mobility tasks performed by persons with paraplegia are wheelchair propulsion and wheelchair transfers. Several investigators have examined upper extremity kinematics (joint motions) kinetics (joint forces and torques), and muscle activity as determined by electromyography (EMG) among individuals with SCI during wheelchair propulsion. Comparatively few studies have addressed wheelchair transfers none of which offer an integrated kinematic, kinetic and EMG approach to simultaneously examine joint angles, moments and muscle activity.

Methods:

Using Vicon motion analysis technology, we propose a laboratory-based randomized evaluation of five vehicle transfer approaches: unassisted manual transfer, standard transfer board, Glide n'Go, Easy Reach lift, and Ryno lift. The selected commercially-available products represent the range of assistive technologies presently available for this task.

A sample of 58 veterans with paraplegia, who use a manual wheelchair for mobility, will be recruited to participate in this study. Subjects will be recruited from the Tampa VA Hospital by means of poster advertisement. Participants will complete data collection activities during one four-hour session, for which they will be compensated. Subjects will be asked to perform a series of five randomized wheelchair-to-vehicle transfer tasks. Vicon markers placed on the participant's body will capture positional data. Dynamic external loads exerted during the transfer tasks will be measured using AMTI MC3A tri-axial load cells strategically mounted in a vehicle mock-up. EMG will be recorded bilaterally for major muscle groups. Participants will complete subjective rating scales upon completion of each of the transfers.

The results of this study will be used to develop a clinical algorithm to assist clinicians with the selection of the most appropriate assistive technology for persons with disabilities who use a manual wheelchair for mobility. This algorithm will facilitate the individualized selection of assistive technologies that minimize risk for injury and maximize patient compliance, comfort, and satisfaction. The ultimate goal of this program of research is to (1) promote successful adaptation to aging with a disability, (2) reduce morbidity and mortality associated with wheelchair use, (3) enhance health-related quality of life, patient freedom, function, independence, and confidence, and (4) reduce healthcare utilization and associated costs.

ELIGIBILITY:
Inclusion Criteria:

* level of SCI will be limited to ASIA A classification at T2 through L5 level to standardize physical capabilities,
* SCI for at least 2 years (neurologically stable,
* use rigid manual wheelchair as a primary means of mobility,
* able to self-propel wheelchair,
* able to independently transfer between wheelchair and vehicle,
* between the ages of 18-65,
* living in the community within 100 miles of the Tampa VA hospital,
* able to follow simple instructions,
* free from acute upper extremity injury for at least six months (determined by chart review) to minimize risk of injury during task performance,
* comparable bilateral functional range of motion and strength of the shoulders, elbows and wrists (determined by physical evaluation) to minimize risk of injury during task performance.

Exclusion Criteria:

Candidates who present:

* progressive disease (e.g. spinal tumor),
* extended bedrest for more than 30 days,
* ventilator-dependent,
* any cardiac or respiratory condition that would limit subject's physical performance,
* unstable medical conditions,
* use of power wheelchair or scooter as primary means of mobility,
* pregnancy,
* clinical evidence of severe musculoskeletal disorders of the upper extremity will be precluded from participating in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A sample of 58 veterans with paraplegia who use a rigid manual wheelchair will be recruited to participate in this study.
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2010-01; Primary Completion 2011-03 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John D Lloyd, PhD BS, Principal Investigator — James A. Haley Veterans' Hospital
Locations (1):
- James A. Haley Veterans' Hospital, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Although 10 individuals signed ICs, 4 actually actively participated in the study as one was dropped due to an unrelated injury.
Groups:
- Wheelchair Transfer Interventions: 5 persons with SCI were recruited and provided informed consent. Four completed the protocol. One was dropped due to an unrelated injury to the subjects hand at his home.
Period: Overall Study
Arm/Group | Wheelchair Transfer Interventions
Started | 5
Completed | 4 (One individual provided consent & was dropped due to an unrelated injury to his hand at his home.)
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: One individual was enrolled in the study but withdrew due to an adverse event (hand injury UNRELATED to the study).
Groups:
- Wheelchair Transfer Interventions: Persons with SCI who evaluated wheelchair transfer interventions
Arm/Group | Wheelchair Transfer Interventions
Number analyzed (Participants) | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.8 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 5

OUTCOME MEASURES:

1. Primary Outcome: Shoulder Force
Description: measurement of applied shoulder force during wheelchair transfers
Time Frame: None reported - verifiable data is not available for any of the participants
Population: As of the November 2012 update to the IRB, there were no findings at that point. At this time, verifiable data is not available for any of the participants.
Groups:
- Glide n' Go; Standard Transfer Board: As of the November 2012 update to the IRB, 4 individuals were reported to actively take part in the study, but verifiable data is not available for any of the participants.
- Easy Reach Lift; Ryno Lift; Unassisted Manual Transfer: As of the November 2012 update to the IRB, 4 individuals were reported to actively take part in the study but verifiable data is not available for any of the participants.
Arm/Group | Glide n' Go | Standard Transfer Board | Easy Reach Lift | Ryno Lift | Unassisted Manual Transfer
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Groups:
- Group 1: persons with SCI
Arm/Group | Group 1
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 1/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=5)
Hand injury (Musculoskeletal and connective tissue disorders) | 1 (1) — UNRELATED hand injury to the subject while he was at his home

LIMITATIONS AND CAVEATS:
PI has left facility. This study did not yield usable results due to staffing, contracting issues. Although 10 individuals signed ICs, 4 actually actively participated in the study and verifiable data is not available for any of the participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes